CLINICAL TRIAL: NCT01074320
Title: Measuring Musculoskeletal Symptoms in Patients Receiving Aromatase Inhibitors
Acronym: AIMS
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 03918-09
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; aromatase inhibitors; musculoskeletal symptoms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients on AIs: Breast cancer patients beginning Aromatase Inhibitor therapy
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — Observational study

SUMMARY:
Current guidelines recommend endocrine treatment with aromatase inhibitors (AIs) in post-menopausal women with hormone receptor-positive breast cancer. Musculoskeletal symptoms are commonly reported with AI treatment,however, we do not have consistent methods to measure these symptoms prospectively. This gap in our knowledge inhibits the ability to test and develop treatments for AI-associated musculoskeletal symptoms. This pilot study will evaluate functional tests and standardized instruments for their ability to prospectively assess musculoskeletal symptoms in women being treated with AIs for breast cancer.

DETAILED DESCRIPTION:
Specific Aims: 1) identify a core set of instruments for measuring musculoskeletal symptoms, 2) model the time course and predictors of change in musculoskeletal symptoms, 3) explore the effect of musculoskeletal symptoms on adherence to AIs in women during the first 6 months of AI treatment.

Methods: We will prospectively assess musculoskeletal symptoms due to treatment with aromatase inhibitors. Post-menopausal women beginning AI treatment for hormone responsive breast cancer will be invited to join this study.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage I - IIIa invasive breast cancer,
* Hormone-receptor positive cancer (either ER+ or PR+ or both),
* Prescribed and have agreed to take exemestane, anastrazole or letrozole,
* Have completed initial treatment of surgery, RT, and/or chemotherapy,
* Are post-menopausal,
* No previous history of aromatase inhibitor therapy for invasive breast cancer,
* Have signed the consent form.

Exclusion Criteria:

* History of rheumatoid arthritis,
* Unable to read or understand English,
* History of psychiatric disability affecting informed consent or compliance with study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-menopausal breast cancer patients receiving aromatase inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Identify a core set of instruments for measuring musculoskeletal symptoms | 09/2011

SECONDARY OUTCOMES:
Model the time course and predictors of change in musculoskeletal symptoms | 09/2011
Explore the effects of musculoskeletal symptoms on adherence to AIs in women during the first 6 months of AI treatment | 09/2011

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Swenson, RN, PhD, Principal Investigator — HealthPartners Institute
Locations (2):
- United States (2):
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota

REFERENCES:
- [Result] Swenson KK, Nissen MJ, Henly SJ, Maybon L, Pupkes J, Zwicky K, Tsai ML, Shapiro AC. Identification of tools to measure changes in musculoskeletal symptoms and physical functioning in women with breast cancer receiving aromatase inhibitors. Oncol Nurs Forum. 2013 Nov;40(6):549-57. doi: 10.1188/13.ONF.549-557. PMID 24161633